CLINICAL TRIAL: NCT02551952
Title: Digital Game MentalPlus®: A Scale to Evaluate on Perioperative Cognitive Function: Content Analysis, Internal Consistency, Convergent Validity and Clinical Validation of the Diagnostic Test
Brief Title: Digital Game: A Scale to Evaluate the Perioperative Cognitive Function
Acronym: MentalPlus®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); University of Copenhagen (Other); Harvard Medical School (HMS and HSDM) (Other); Max Planck Institute for Human Development (Other)
Responsible Party: Principal Investigator, Livia Stocco Sanches Valentin, Ph.D., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Interventional Study Design
Record Dates: First submitted 2015-08-31; First posted 2015-09-16 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cognition Disorders; Impaired Cognition; Self-Assessment
Keywords: Games; Cognitive Tests; General Anesthesia; Surgery
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Intervention Model Description: The study was conceived as a randomized, double-blind exploratory trial. It received the approval of the Ethics Committee for Research Project Analysis (CAPPesq) of the Clinical Board, Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC-FMUSP).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization was performed using the website http://www.randomizer.org/form.htm, recorded on paper and stored in sealed opaque envelopes to be opened in the study room where volunteers would play the video game. The health professionals responsible for the game application were aware of the MentalPlus® game version arm just after openness of the envelopes. However, patients, neuropsychologists, and outcome assessors involved in the the study was kept blinded to the stratification group to which each patient belonged. The study groups were identified only after the evaluation of all patients and statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MentalPlus® PILOT-I (Experimental): This preliminary group will be submitted to the digital game MentalPlus®, also be the submitted to fMRI before and after surgery. The results of standardized tests and the data of the MentalPlus® of patients undergoing surgery will be compared with the results of the same tests and the data of the MentalPlus® of healthy volunteers with similar characteristics regarding the variables age and education.
  Interventions: Device: MentalPlus®
- MentalPlus® PILOT-II (Experimental): This preliminary group will be of healthy volunteers submitted to the digital game MentalPlus®. The results of standardized tests and the data of the MentalPlus® of volunteers will be compared with the results of tests of patients undergoing surgery and the data of the MentalPlus®.
  Interventions: Device: MentalPlus®
- Group I: MentalPlus® (Active Comparator): Evaluated with neuropsychological tests and MentalPlus® before surgery. After surgery, from the 3rd postoperative day a tablet will be use with MentalPlus® in 7 versions for cognitive training during 7 days (7 versions with interfaces adapted for ages up to 20 years and 7 versions for ages over it).
  Interventions: Device: MentalPlus®
- Group II: MentalPlus® (Sham Comparator): Ratings with neuropsychological testing and evaluation with MentalPlus® before surgery will be realized. After surgery, from the 3rd postoperative day a tablet will be use for entertainment with short films (20 minutes) for use in the placebo effect of digital game MentalPlus® this group also will be submitted to fMRI before and after surgery. (With the intention to respond to the specificity of findings in relation to the control for active placebo effect)
  Interventions: Device: MentalPlus®

INTERVENTIONS:
Device: MentalPlus® — Validate the MentalPlus® digital game as neuropsychological test of cognitive assessment pre and postoperative on study the internal consistency and validity of content and construct (convergent) MentalPlus® of the evaluated patients. Study the influence of age, gender and level of education of surgical patients in performance for the use of electronic devices (laptop, tablet, mobile) and digital games. Investigate the rehabilitation capacity of cognitive functions after training sessions with MentalPlus® game. Evaluate the effect of training with MentalPlus® game in brain networks involved in executive function, memory and attention by means of fMRI this is a brain imaging study.
  Other Names: Brazilian National Library Foundation nº 663707

SUMMARY:
INTRODUCTION: Cognitive dysfunction is a frequent adverse event in the postoperative period, especially in elderly patients. The tests commonly used for the detection of postoperative cognitive dysfunction are time-consuming and with variable sensitivity and specificity and difficult routine use. Applying a difficult battery of cognitive tests decreases the viability of adopting measures to increase preoperative cognitive reserve and methods for prevention, diagnosis and rehabilitation of cases of Postoperative Cognitive Dysfunction (POCD), it is desirable to search for alternative methods diagnoses.

DETAILED DESCRIPTION:
Thinking about this concern, the investigators created a digital game to assess quickly and funny the cognitive functions (memory; attention and executive). The investigators know that digital games have potential neuromodulator effect and have been used as an alternative to the psychotherapeutic treatment and rehabilitation of cognitive skills. However, the experience with these games to assess the integrity of perioperative neuropsychological functions is still scarce. It is hypothesized that a digital game can replace the commonly used neuropsychological tests for detecting postoperative cognitive dysfunction. The aim of this study is to validate a specific digital game (MentalPlus®) for cognitive assessment and evaluation of its use for detecting of postoperative cognitive dysfunction.

METHODS: The participants will be studied over 20 years old, literate, of both genders and candidates for surgery under general anesthesia in the Clinics Hospital of the Faculty of Medicine, University of São Paulo. Will also be applied neuropsychological tests to evaluate memory, attention, and executive functions as well as another tests to assess specifics contents useful to describe the sample and research' results. The tests applied will be on specific data set. In another study the investigators will include volunteers to assess short and long term memory Verbal Learnings Test (VLT), visual memory with Recognition Memory Test (TEM-R), to executive functions with STROOP Test and the selective and alternating attention with Trail Making Test (TMT-A / B). For Quality of Life the investigators will use the Patient Health Questionnaire (PHQ-9) and Beck Depression Inventory (BDI-II) and Beck Anxiety Inventory (BAI) to assess depressive and anxiety symptoms, beyond of the MentalPlus®. In a third project the investigators will use functional magnetic resonance imaging (fMRI) to assess the association between brain response and cognitive training by MentalPlus®. Reliability analysis will be performed and the validity of the digital game will be assessed in terms of evaluation of cognitive functions in a fun and practical way and this may provide health professionals, including anesthesiologists and surgeons with a new method for neuropsychological evaluation.

Detail description about the neuropsychological tests and scales: Sociodemographic data will be analyzed including education, marital status, occupation, and current medication. Signs and symptoms of depression will be assess preoperatively using the Beck Depression Inventory (BDI), for screening on global cognitive will be use Telephone Interview for Cognitive Status (TICS), will be use the Verbal Learning Test (VLT) for long-term memory and the Recognition Memory Test (TEM-R) for visual memory, the Symbol Digit Modified Test (SDMT) will be use to assess short-term memory, visual search skill and attention, STROOP Test will be assess the selective attention, inhibitory ability and mental flexibility that are constructs of executive function and the Trail Making Test (TMT) for the assessment of selective and alternating attention.

Beck Depression Inventory (BDI), which consists of 21 questions that explore depressive symptoms on a scale of 0 to 4, where zero represents no symptoms and four is the maximum symptomatology. A total of 14 points will be consider indicative of the presence of moderate depressive symptoms22.

Patient Questionnaire health (PHQ-9), this questionnaire about the health of the patient is an instrument with 9 questions. Each question has 4 possible responses: 0 (no day), 1 (several days), 2 (more than half days), and 3 (nearly every day). The PHQ-9 can be interpreted in three ways: 10 in the form of algorithm, identifying individuals with a major depressive episode and tracking probable cases of major depressive disorder; 20 as a continuous measure, with scores between 0 and 27 points, being able to assess levels of depressive symptoms through the cut- points 5, 10, 15 and 20 points = mild depression, moderate, severe and serious; 30 as continuous measurements with scores between 0 and 27 points, classifying the individuals dichotomous through the use of a single cutting point (typically ≥10).

The Telephone Interview for Cognitive Status (TICS) will be use as a standardized test to assess neuropsychological functioning when assessing cognitive skills. This test can be used when screening personally is impractical or when patients are unable to attend the clinic. This test consists of a structured interview with 11 items that assess the skills of spatial and temporal orientation, mental control, memory, general information, language and calculations.

Memory will be assessed using the Verbal Learning Test (VLT) this test consists of a list of words. A list of 15 words is presented and must to be stored and recalled in three successive attempts (VLT / A-B-C), with delayed recall after 25 minutes (VLT-Delay). Rate is the number of words recalled and the number of errors for each presentation. The VLT evaluates the modalities of memory immediate, consolidated and long-term. This instrument will be held in two stages: pre-operative at the time of 1st evaluation before surgery and postoperatively in the second and final assessment between day 10 and 15 postoperatively.

The Recognition Memory Test (TEM-R) consists of storing pictures and words to further identify remembered stimuli. For the stimulus responses can be presented to the subject in graphic form (figures) or written (words). This instrument will be held in two stages: pre-operative at the time of 1st evaluation before surgery and postoperatively in the second and final assessment between day 10 and 15 postoperatively.

The Symbol Digit Modified Test (SDMT) will be applied for the evaluation of short-term memory, visual search skill and attention. This is a graphical task where the individual has to fill in symbols exemplified in the spaces below the corresponding number within 180 seconds. The result is measured as the number of symbols drawn and the number of errors.

Attention will be assessed by STROOP Test, which consists in presenting three paper sheets to the subject. The first one, the patient should verbalize the names of colors printed in black ink. In the second, verbalization is made of color are filled rectangles, the same provision of the words of the previous slide. The third blade consist in verbalize colors printed over the written word. Evaluates selective attention, inhibitory ability and mental flexibility that are constructs of executive function. Scores obtained include the number of words (Word task), number of bar colors (Color), and number of color words (Color-Word) completed within a set time, or as noted above, the amount of time required to complete each of the tasks. We will consider the number of errors as well.

Attention will also be evaluated using the Trail Making Test (TMT) for the assessment of selective and alternating attention. In part A of the test, the subject must draw lines connecting consecutively numbered circles. In part B, the subject must draw lines connecting circles alternately with letters and numbers in a sequence. The result is measured as time and trail errors. The Attention function will be examined with Trail Making Test (TMT). This test consists of two parts. In Part A, the subject must draw lines connecting consecutively numbered circles. In Part B, the subject must draw lines alternately connecting circles with letters and numbers in a sequence. The test involves addition of alternate and selective attention, visual screening and complex manual dexterity (Part A) and executive processes (Part B). Among the executive procedures, the inhibitory ability and cognitive alternating seem to be those most required in completing the task. They are valued the time spent and the number of errors in each of. These instrument will be held in two stages: pre-operative at the time of 1st evaluation before surgery and postoperatively in the second and final assessment between day 10 and 15 postoperatively.

About the scale for validation: the study will be guided on the validation of a digital game MentalPlus® in the form of scale to assess the neuropsychological functions: attention, memory, and executive. This scale will be measured with scores ranging between 0 and 20 to corrects and errors. Attention function: 0 (zero) corresponds to much trouble (too many errors); twenty (20) corresponds full capacity (correct total).

For the executive function will be assessed: capacity of resistance for distractor factor being measured by how much that person touches the tablet's screen in order to demonstrate the failure of inhibitory control of the actions. Scores between 0 and 20 where 0 (zero) means great inhibitory control up to twenty (20) total inability to inhibitory control.

For the memory function will be assessed the long-term memory, working memory and short-term visual memory. The scores for this function range from 0 to 20, with 0 (zero) total memorizing inability to long-term task and twenty (20) total long-term storage capacity evaluated after 25 minutes of exposure of the figures to be memorized. For the working memory will be exposed 7 icons to be mentioned over the next five minutes of exposure. Seven (7)= good ability to manipulate information in short-term time and 0 (zero) inability to store and manipulate information in short time.

ELIGIBILITY:
Inclusion Criteria:

* Be a candidate for elective surgery small and medium-sized under general anesthesia for any surgical specialty. Have at least nine years of schooling or more, have between 20 and 40 years and want to participate in the research of their own free will.
* diagnosis of Hypertension of Pressure Normal (HPN), the absence of malignancy, well-controlled clinical comorbidities (hypertension, diabetes mellitus, hormonal disorders, etc.) with predictive tools of post surgery results: tap test, lumbar infusion test, and continuous 72-hours external lumbar drainage and pressure monitoring.

Exclusion Criteria:

* Provide a history of psychiatric disorders and dementias that affect cognition, lack of knowledge of the Portuguese language, use metal clips or cardiac pacemaker that preclude the examination by Functional Magnetic Resonance Imaging.
* diagnosis of secondary HPN, inability to walk, malignancy, clinical comorbidities uncontrolled presenting a history of psychiatric disorders and dementias that affect cognition, for instance Alzheimer's Dementia, lack of knowledge of the Portuguese language, use metal clips or marked heart step, which makes the examination by Functional Magnetic Resonance Imaging no functionality.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Measures of cognitive functions: executive, memory and attention on the MentalPlus® Scale | 20 minutes
  Scores range from 0 [Not improved] to 10 [fully improved] at cognitive functions memory, attention and executive after training with MentalPlus® Scale and compared with neuropsychological tests validated and standardised to the global population.

SECONDARY OUTCOMES:
Change From Baseline in Neuropsychological Scores on the MentalPlus® Scale for memory, attention and executive function at 20 days. | 20 days
  Scores range from 0 [Not improved] to 10 [fully improved] at cognitive functions memory, attention and executive after training with MentalPlus® Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lívia SS Valentin, Ph.D., Principal Investigator — Faculty of Medicine of the University of Sao Paulo
Locations (1):
- Livia Stocco Sanches Valentin, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hudetz JA, Iqbal Z, Gandhi SD, Patterson KM, Hyde TF, Reddy DM, Hudetz AG, Warltier DC. Postoperative cognitive dysfunction in older patients with a history of alcohol abuse. Anesthesiology. 2007 Mar;106(3):423-30. doi: 10.1097/00000542-200703000-00005. PMID 17325499
- [Result] Youngblom E, DePalma G, Sands L, Leung J. The temporal relationship between early postoperative delirium and postoperative cognitive dysfunction in older patients: a prospective cohort study. Can J Anaesth. 2014 Dec;61(12):1084-92. doi: 10.1007/s12630-014-0242-6. Epub 2014 Oct 7. PMID 25287962
- [Result] Boos GL, Soares LF, Oliveira Filho GR. [Postoperative cognitive dysfunction: prevalence and associated factors.]. Rev Bras Anestesiol. 2005 Oct;55(5):517-24. doi: 10.1590/s0034-70942005000500006. Portuguese. PMID 19468642
- [Result] Burkhart CS, Steiner LA. Can postoperative cognitive dysfunction be avoided? Hosp Pract (1995). 2012 Feb;40(1):214-23. doi: 10.3810/hp.2012.02.962. PMID 22406897
- [Result] Damuleviciene G, Lesauskaite V, Macijauskiene J. [Postoperative cognitive dysfunction of older surgical patients]. Medicina (Kaunas). 2010;46(3):169-75. Lithuanian. PMID 20516755
- [Result] Blumberg FC, Fisch SM. Introduction: digital games as a context for cognitive development, learning, and developmental research. New Dir Child Adolesc Dev. 2013 Spring;2013(139):1-9. doi: 10.1002/cad.20026. PMID 23483688
- [Result] Green CS, Bavelier D. Learning, attentional control, and action video games. Curr Biol. 2012 Mar 20;22(6):R197-206. doi: 10.1016/j.cub.2012.02.012. PMID 22440805
- [Result] Fernandez-Aranda F, Jimenez-Murcia S, Santamaria JJ, Gunnard K, Soto A, Kalapanidas E, Bults RG, Davarakis C, Ganchev T, Granero R, Konstantas D, Kostoulas TP, Lam T, Lucas M, Masuet-Aumatell C, Moussa MH, Nielsen J, Penelo E. Video games as a complementary therapy tool in mental disorders: PlayMancer, a European multicentre study. J Ment Health. 2012 Aug;21(4):364-74. doi: 10.3109/09638237.2012.664302. Epub 2012 May 1. PMID 22548300
- [Result] Kuhn S, Lorenz R, Banaschewski T, Barker GJ, Buchel C, Conrod PJ, Flor H, Garavan H, Ittermann B, Loth E, Mann K, Nees F, Artiges E, Paus T, Rietschel M, Smolka MN, Strohle A, Walaszek B, Schumann G, Heinz A, Gallinat J; IMAGEN Consortium. Positive association of video game playing with left frontal cortical thickness in adolescents. PLoS One. 2014 Mar 14;9(3):e91506. doi: 10.1371/journal.pone.0091506. eCollection 2014. PMID 24633348
- [Result] Kuhn S, Gleich T, Lorenz RC, Lindenberger U, Gallinat J. Playing Super Mario induces structural brain plasticity: gray matter changes resulting from training with a commercial video game. Mol Psychiatry. 2014 Feb;19(2):265-71. doi: 10.1038/mp.2013.120. Epub 2013 Oct 29. PMID 24166407
- [Result] Anguera JA, Boccanfuso J, Rintoul JL, Al-Hashimi O, Faraji F, Janowich J, Kong E, Larraburo Y, Rolle C, Johnston E, Gazzaley A. Video game training enhances cognitive control in older adults. Nature. 2013 Sep 5;501(7465):97-101. doi: 10.1038/nature12486. PMID 24005416
- [Result] Rosser JC Jr, Lynch PJ, Cuddihy L, Gentile DA, Klonsky J, Merrell R. The impact of video games on training surgeons in the 21st century. Arch Surg. 2007 Feb;142(2):181-6; discusssion 186. doi: 10.1001/archsurg.142.2.181. PMID 17309970
- [Result] Patel A, Schieble T, Davidson M, Tran MC, Schoenberg C, Delphin E, Bennett H. Distraction with a hand-held video game reduces pediatric preoperative anxiety. Paediatr Anaesth. 2006 Oct;16(10):1019-27. doi: 10.1111/j.1460-9592.2006.01914.x. PMID 16972829
- [Result] Russoniello CV, O'Brien K, Parks JM. EEG, HRV and Psychological Correlates while Playing Bejeweled II: A Randomized Controlled Study. Stud Health Technol Inform. 2009;144:189-92. PMID 19592761
- [Result] Saleem M, Anderson CA, Gentile DA. Effects of Prosocial, Neutral, and Violent Video Games on Children's Helpful and Hurtful Behaviors. Aggress Behav. 2012 Jul-Aug;38(4):281-7. doi: 10.1002/ab.21428. PMID 25363697
- [Result] Montag C, Weber B, Trautner P, Newport B, Markett S, Walter NT, Felten A, Reuter M. Does excessive play of violent first-person-shooter-video-games dampen brain activity in response to emotional stimuli? Biol Psychol. 2012 Jan;89(1):107-11. doi: 10.1016/j.biopsycho.2011.09.014. Epub 2011 Oct 5. PMID 21982747
- [Result] Gentile DA, Choo H, Liau A, Sim T, Li D, Fung D, Khoo A. Pathological video game use among youths: a two-year longitudinal study. Pediatrics. 2011 Feb;127(2):e319-29. doi: 10.1542/peds.2010-1353. Epub 2011 Jan 17. PMID 21242221
- [Result] Bavelier D, Green CS, Pouget A, Schrater P. Brain plasticity through the life span: learning to learn and action video games. Annu Rev Neurosci. 2012;35:391-416. doi: 10.1146/annurev-neuro-060909-152832. PMID 22715883
- [Result] Oei AC, Patterson MD. Enhancing cognition with video games: a multiple game training study. PLoS One. 2013;8(3):e58546. doi: 10.1371/journal.pone.0058546. Epub 2013 Mar 13. PMID 23516504
- [Result] Boot WR, Blakely DP, Simons DJ. Do action video games improve perception and cognition? Front Psychol. 2011 Sep 13;2:226. doi: 10.3389/fpsyg.2011.00226. eCollection 2011. PMID 21949513
- [Result] Hommel B, Colzato LS. Games with(Out) Frontiers: Toward an Integrated Science of Human Cognition. Front Psychol. 2010 Mar 8;1:2. doi: 10.3389/fpsyg.2010.00002. eCollection 2010. No abstract available. PMID 21833185
- [Result] Merabet LB, Connors EC, Halko MA, Sanchez J. Teaching the blind to find their way by playing video games. PLoS One. 2012;7(9):e44958. doi: 10.1371/journal.pone.0044958. Epub 2012 Sep 19. PMID 23028703
- [Result] Thompson JJ, Blair MR, Chen L, Henrey AJ. Video game telemetry as a critical tool in the study of complex skill learning. PLoS One. 2013 Sep 18;8(9):e75129. doi: 10.1371/journal.pone.0075129. eCollection 2013. PMID 24058656
- [Result] Sanchez CA. Enhancing visuospatial performance through video game training to increase learning in visuospatial science domains. Psychon Bull Rev. 2012 Feb;19(1):58-65. doi: 10.3758/s13423-011-0177-7. PMID 22037919
- [Result] Mathewson KE, Basak C, Maclin EL, Low KA, Boot WR, Kramer AF, Fabiani M, Gratton G. Different slopes for different folks: alpha and delta EEG power predict subsequent video game learning rate and improvements in cognitive control tasks. Psychophysiology. 2012 Dec;49(12):1558-70. doi: 10.1111/j.1469-8986.2012.01474.x. Epub 2012 Oct 23. PMID 23095124
- [Result] Maclin EL, Mathewson KE, Low KA, Boot WR, Kramer AF, Fabiani M, Gratton G. Learning to multitask: effects of video game practice on electrophysiological indices of attention and resource allocation. Psychophysiology. 2011 Sep;48(9):1173-83. doi: 10.1111/j.1469-8986.2011.01189.x. Epub 2011 Mar 9. PMID 21388396
- [Result] Cardoso-Leite P, Bavelier D. Video game play, attention, and learning: how to shape the development of attention and influence learning? Curr Opin Neurol. 2014 Apr;27(2):185-91. doi: 10.1097/WCO.0000000000000077. PMID 24553464
- [Result] Deveau J, Lovcik G, Seitz AR. Broad-based visual benefits from training with an integrated perceptual-learning video game. Vision Res. 2014 Jun;99:134-40. doi: 10.1016/j.visres.2013.12.015. Epub 2014 Jan 6. PMID 24406157
- [Result] Valentin LSS, Valentin TSS, Carmona MJC, Aguilar G, Pires VY, Garcia RC, et al. Digital Game Test Neuropsychology. Fundação Biblioteca Nacional. 2014.
- [Result] Valentin LSS, Valentin TSS, Carmona MJC, Garcia RC, Correa RD, Gondim GB, et al. Mental Plus. INPI - Instituto Nacional da Propriedade Intelectual. 2014.
- [Result] Tang J, Eckenhoff MF, Eckenhoff RG. Anesthesia and the old brain. Anesth Analg. 2010 Feb 1;110(2):421-6. doi: 10.1213/ANE.0b013e3181b80939. Epub 2009 Oct 9. PMID 19820235
- [Result] Asilioglu K, Celik SS. The effect of preoperative education on anxiety of open cardiac surgery patients. Patient Educ Couns. 2004 Apr;53(1):65-70. doi: 10.1016/S0738-3991(03)00117-4. PMID 15062906
- [Result] Naismith SL, Longley WA, Scott EM, Hickie IB. Disability in major depression related to self-rated and objectively-measured cognitive deficits: a preliminary study. BMC Psychiatry. 2007 Jul 17;7:32. doi: 10.1186/1471-244X-7-32. PMID 17634111
- [Result] Postler A, Neidel J, Gunther KP, Kirschner S. Incidence of early postoperative cognitive dysfunction and other adverse events in elderly patients undergoing elective total hip replacement (THR). Arch Gerontol Geriatr. 2011 Nov-Dec;53(3):328-33. doi: 10.1016/j.archger.2010.12.010. Epub 2011 Feb 1. PMID 21288579
- [Result] Koster S, Hensens AG, van der Palen J. The long-term cognitive and functional outcomes of postoperative delirium after cardiac surgery. Ann Thorac Surg. 2009 May;87(5):1469-74. doi: 10.1016/j.athoracsur.2009.02.080. PMID 19379886
- [Result] Schmiedek F, Lovden M, Lindenberger U. Hundred Days of Cognitive Training Enhance Broad Cognitive Abilities in Adulthood: Findings from the COGITO Study. Front Aging Neurosci. 2010 Jul 13;2:27. doi: 10.3389/fnagi.2010.00027. eCollection 2010. PMID 20725526
- [Result] Mori E, Ishikawa M, Kato T, Kazui H, Miyake H, Miyajima M, Nakajima M, Hashimoto M, Kuriyama N, Tokuda T, Ishii K, Kaijima M, Hirata Y, Saito M, Arai H; Japanese Society of Normal Pressure Hydrocephalus. Guidelines for management of idiopathic normal pressure hydrocephalus: second edition. Neurol Med Chir (Tokyo). 2012;52(11):775-809. doi: 10.2176/nmc.52.775. PMID 23183074
- [Result] Shprecher D, Schwalb J, Kurlan R. Normal pressure hydrocephalus: diagnosis and treatment. Curr Neurol Neurosci Rep. 2008 Sep;8(5):371-6. doi: 10.1007/s11910-008-0058-2. PMID 18713572
- [Result] Vieira G, Amaro E Jr, Baccala LA. Local sparse component analysis for blind source separation: an application to resting state FMRI. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:5611-4. doi: 10.1109/EMBC.2014.6944899. PMID 25571267
- [Result] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Result] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Result] Beck AT SR. Beck depression Inventory. manual. San Antonio: Psychology Corporation. 1993.
- [Result] Baccaro A, Segre A, Wang YP, Brunoni AR, Santos IS, Lotufo PA, Bensenor IM, Goulart AC. Validation of the Brazilian-Portuguese version of the Modified Telephone Interview for cognitive status among stroke patients. Geriatr Gerontol Int. 2015 Sep;15(9):1118-26. doi: 10.1111/ggi.12409. Epub 2014 Nov 19. PMID 25407304
- [Result] Cavaco S, Goncalves A, Pinto C, Almeida E, Gomes F, Moreira I, Fernandes J, Teixeira-Pinto A. Auditory Verbal Learning Test in a Large Nonclinical Portuguese Population. Appl Neuropsychol Adult. 2015;22(5):321-31. doi: 10.1080/23279095.2014.927767. Epub 2015 Jan 12. PMID 25580839
- [Result] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086